CLINICAL TRIAL: NCT03375671
Title: Rapid Agitation Control With Ketamine in the Emergency Department (RACKED): a Randomized Controlled Trial
Brief Title: Rapid Agitation Control With Ketamine in the Emergency Department
Acronym: RACKED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Barbic (Other)
Collaborators: St Paul's Emergency Department Research Fund (Unknown); Centre for Health Evaluation and Outcome Sciences (CHÉOS) (Unknown)
Responsible Party: Sponsor-Investigator, David Barbic, Clinical Assistant Professor, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H17-00571
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Violent Aggressive Behavior; Ketamine
Keywords: ketamine; aggressive behaviour; midazolam; haloperidol; emergency department
MeSH Terms: conditions — Aggression; Emergencies | interventions — Ketamine; Midazolam; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Single administration of Ketalar® (ketamine hydrochloride injection, USP); 5 mg/kg, IM
  Interventions: Drug: Ketalar
- Midazolam + haloperidol (Active Comparator): Single administration of combination of: Midazolam injection (5 mg, IM) and haloperidol injection (5mg, IM)
  Interventions: Drug: Midazolam injection; Drug: Haloperidol

INTERVENTIONS:
Drug: Ketalar — single administration of 5 mg/kg, IM
  Other Names: ketamine
  Arms: Ketamine
Drug: Midazolam injection — single administration of 5 mg, IM
  Arms: Midazolam + haloperidol
Drug: Haloperidol — single administration of 5 mg, IM
  Arms: Midazolam + haloperidol

SUMMARY:
Compare intramuscular (IM) ketamine to a combination of IM midazolam and haloperidol with regards to the time required for adequate behavioral control, in minutes, in patients presenting to the emergency department with psychomotor agitation and violent behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 - 60 years inclusively;
2. Patients presenting to the emergency department with psychomotor agitation or violent behaviour (RASS score > +3).

Exclusion Criteria:

1. Less than 19 years of age;
2. Greater than 60 years of age;
3. Previous participation in this study;
4. Women suspected or known to be pregnant or breastfeeding;
5. Previous known hypersensitivity, intolerance or allergy to ketamine, midazolam or haloperidol or their components.
6. Subjects who are in comatose states or have CNS depression due to alcohol or are taking other depressant drugs.
7. Subjects with severe depressive states, spastic diseases and in Parkinson's syndrome, except in the case of dyskinesias due to levodopa treatment.
8. Senile patients with pre-existing Parkinson-like symptoms.
9. Subjects with a history of cerebrovascular accident
10. Subjects in whom a significant elevation of blood pressure would constitute a serious hazard, such as patients with significant hypertension
11. Subjects with severe cardiac decompensation
12. Subjects who intend to have surgery of the pharynx, larynx, or bronchial tree unless adequate muscle relaxants are used
13. Subjects with acute pulmonary insufficiency
14. Subjects with severe chronic obstructive pulmonary disease
15. Subjects with acute narrow angle glaucoma

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Time from first IM medication administration to adequate sedation which is defined as RASS less than or equal to -1. | 1 day
  Measured using Richmond Agitation Sedation Scale (RASS) in each arm

SECONDARY OUTCOMES:
Percentage participants with adverse events in each arm | up to 4 days
  measured by AE collection in each arm
Percentage of participants in each arm requiring rescue medications between 5 and 30 minutes (at 5 minutes interval) after study medication(s) administration by count. | 1 day
  measured by rescue medication administration
Percentage of participants in each arm experiencing sedation outcomes as defined by the TROOPS criteria | 1 day
  measured using Tracking and Reporting Outcomes of Procedural Sedation (TROOPS) criteria
Percentage of participants with neuroleptic malignant syndrome events within 24 hours of enrollment of each arm. | 1 day
  measured by occurrence of neuroleptic malignant syndrome
Percentage of participants experiencing pre-hospital use of force by police in this participant population, by number and type of restraint. | 1 day
  measured by police account at study enrollment
Participant experience survey outcomes. | 1 day
  measured using Participant Experience Survey
Study Nurse Experience survey outcomes. | 1 day
  measured using Study Nurse Experience Survey
Effectiveness of Blinding survey outcomes | 1 day
  measured using Effectiveness of Study Drug Blinding Survey

CONTACTS AND LOCATIONS:
Overall Officials: David Barbic, MD MSc FRCPC,, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital Emergency Department, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barbic D, Andolfatto G, Grunau B, Scheuermeyer FX, MacEwan W, Honer WG, Wong H, Barbic SP. Rapid agitation control with ketamine in the emergency department (RACKED): a randomized controlled trial protocol. Trials. 2018 Nov 26;19(1):651. doi: 10.1186/s13063-018-2992-x. PMID 30477544